CLINICAL TRIAL: NCT03311477
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of ABBV-399 in Japanese Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics ABBV-399 in Japanese Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-080
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: ABBV-399; Maximum tolerated dose (MTD); Maximally administered dose (MAD); Dose escalation; Pharmacokinetics; Advanced solid tumors; Cancer; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-399 (Experimental): ABBV-399 via intravenous administration at escalating dose levels.
  Interventions: Drug: ABBV-399

INTERVENTIONS:
Drug: ABBV-399 — Intravenous infusion

SUMMARY:
An open-label, dose-escalation study designed to evaluate the safety, pharmacokinetics, and preliminary efficacy of ABBV-399 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant with histologically confirmed advanced solid tumor.
* Participant must have advanced solid tumor that is not amenable to surgical resection or other approved therapeutic options that have demonstrated clinical benefit.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Participant must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Participant has archived diagnostic formalin-fixed paraffin embedded (FFPE) tumor tissue available for analysis.
* Participant has adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

* Participant has received anticancer therapy including chemotherapy, immunotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within a period of 21 days, or herbal therapy within 7 days prior to the first dose of ABBV-399.
* Participant has known uncontrolled metastases to the central nervous system. Participants with brain metastases are eligible after definitive therapy provided they are asymptomatic off systemic steroids and anticonvulsants for at least 2 weeks prior to first dose of ABBV-399.
* Participant has unresolved clinically significant adverse events >= Grade 2 from prior anticancer therapy except for alopecia or anemia.
* Participant has had major surgery within 21 days prior to the first dose of ABBV-399.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t) | Up to 24 months
  AUC (0-t) is defined as area under the concentration versus time curve from time zero (pre-dose) to the time of the last measurable concentration.
Maximum Tolerated Dose (MTD) or maximally administered dose (MAD) for ABBV-399 | Up to 21 days
  MTD/MAD is defined as the highest dose level at which less than 2 of 6 (or < 33% if cohort is expanded beyond 6) participants experience a dose limiting toxicity.
Terminal elimination half life (t1/2) | Up to 24 months
  Terminal elimination half life (t1/2)
Maximum Observed Concentration (Cmax) | Up to 24 months
  Maximum observed concentration (Cmax)
Time to Cmax (Tmax) | Up to 24 months
  Time to Cmax (Tmax)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Time | Up to 24 months
  PFS time is defined as the time from the participant's first dose of ABBV-399 to either the participant's disease progression or death, whichever occurs first.
Objective Response Rate (ORR) | Up to 24 months
  Objective response rate (ORR) is defined as the proportion of participants with a confirmed partial or complete response to the treatment. Evaluation of tumor response is based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of response (DOR) | Up to 24 months
  DOR is defined as the time from the participant's initial objective response to study drug therapy to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (2):
- Japan (2):
  - Shizuoka Cancer Center /ID# 166940, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 166939, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fujiwara Y, Kenmotsu H, Yamamoto N, Shimizu T, Yonemori K, Ocampo C, Parikh A, Okubo S, Fukasawa K, Murakami H. Phase 1 study of telisotuzumab vedotin in Japanese patients with advanced solid tumors. Cancer Med. 2021 Apr;10(7):2350-2358. doi: 10.1002/cam4.3815. Epub 2021 Mar 6. PMID 33675179